CLINICAL TRIAL: NCT04373330
Title: Healthy Living Partnerships for Veterans With Migraine
Acronym: HELP-VM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of Personnel
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: W.G. Bill Hefner Medical Center (U.S. Federal Agency); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB00064225; UL1TR001420 (NIH)
Record Dates: First submitted 2020-04-29; First posted 2020-05-04 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-02

CONDITIONS: Migraine; Migraine Disorders; Migraine With Aura; Migraine Without Aura
MeSH Terms: conditions — Migraine Disorders; Migraine with Aura; Migraine without Aura

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive lifestyle intervention (Experimental): The intensive lifestyle intervention used in HELP PD and that will be used in HELP-VM was a modification of the successful Diabetes Prevention Program (DPP) core curriculum adapted for use in groups. The 16-session core curriculum used in DPP, covering key concepts related to energy balance, nutrition, and physical activity, was expanded to include regular sessions focused on group problem-solving of barriers and issues specific to the members and to incorporate presentations from local community groups on topics relevant to healthy living (exercise resources, etc.) The same intervention will be used in HELP-VM and will target moderate intensity physical activity (goal ≥180 min/wk). A DVD series was developed in HELP PD to standardize this core content, improve fidelity of intervention delivery, and to allow the CHWs to focus on group facilitation and problem-solving. This DVD series will also be used in HELP-VM.
  Interventions: Behavioral: Intensive Lifestyle Intervention
- Medical Treatment as Usual (No Intervention): Subjects randomized to MTAU will be encouraged to continue engaging in medical treatment as per their usual. The MTAU group will complete baseline and 6-month follow-up assessments, and participants will complete daily symptom self-monitoring on the same schedule as HELP-VM participants.

INTERVENTIONS:
Behavioral: Intensive Lifestyle Intervention — There will be 14 sessions delivered over the course of 6 months; materials consist of CHW lesson plans, participant workbooks, and the DVD series. These materials will be adapted for use in HELP-VM and will include information on migraine and its management as well as mental health resources available to Veterans for common illnesses like depression and post-traumatic stress disorder and modifying physical activity recommendations for Veterans with limited mobility.
  Arms: Intensive lifestyle intervention

SUMMARY:
This pilot study, modeled upon the successful and empirically validated HELP Prevent Diabetes Intervention, incorporates a migraine education component describing the links between lifestyle behaviors and migraine activity (e.g., frequency, impairment) into an existing lifestyle intervention used previously for Veterans at risk for developing Type II diabetes. The principal objectives of this research are to assess the feasibility, acceptability (recruitment), engagement (retention, adherence), and promise of implementing the HELP-VM at the Salisbury. To achieve our objectives, the investigators propose to assess the acceptability of HELP-VM by determining our ability to recruit Veterans to participate in the HELP-VM intervention as administered through the existing structure of the Salisbury VAMC's Whole Health Program, to evaluate the feasibility of implementing HELP-VM by assessing Veterans' adherence to HELP-VM and our capacity to retain them in a clinical trial, and to evaluate the promise of HELP-VM by obtaining preliminary data to estimate variances of primary (headache frequency, headache-related impairment) and secondary/exploratory outcome measures (e.g., emotional distress, use of analgesics/opiates, headache self-efficacy, pain catastrophizing) to inform a future, large-scale trial.

DETAILED DESCRIPTION:
Headache disorders such as migraine occur commonly among Veterans and contribute to disability and reduced quality of life. Veterans with migraine are more likely than those without headache to experience medically related discharge/retirement, post-traumatic stress disorder, sleep disturbances, and difficulty reintegrating back into civilian life.

Despite advances in our understanding of migraine, it remains poorly understood and often proves refractory to validated drug and non-drug interventions. Therefore, there is tremendous potential value in pursuing alternate intervention pathways for migraine management. Although empirical support remains limited, engagement in regular exercise routinely is recommended for managing and preventing migraine.

This innovative approach, if successful, could be disseminated rapidly to the VAMC in the United States, thereby making a substantial impact on the public health burden of migraine and other lifestyle related chronic diseases amongst our nation's Veterans. Consistent with the VA's Whole Health Initiative, this HELP-VM approach facilitates and supports Veterans' capacity to take charge of their own health and well-being, and recognizes the many health benefits of reducing sedentary activity for migraine and beyond.

ELIGIBILITY:
Inclusion Criteria:

* Demographics: Community dwelling men and women Veterans (21 years of age and older) of all races/ethnicities seen as patients at the Kernersville Health Care Center.
* Headache Diagnosis, frequency, and chronicity: All participants will be required to have a diagnosis of chronic migraine as per ICHD-IIIβ criteria24. Those with headache frequency ≥ 15 headache days per month for more than three months will be eligible to participate.
* Willingness to Accept Randomization: Prospective participants must be willing to accept randomization to either the intensive lifestyle intervention or the comparison intervention condition.
* Baseline Physician Activity Level: At the time of enrollment, prospective participants must not be participating in a regular physical activity or exercise regimen, and should meet the criteria for "sedentary" (i.e., does not report current engagement in vigorous or moderate activity) on the International Physical Activity Questionnaire Short form (IPAQ-SF).

Exclusion Criteria:

* Other painful conditions: A diagnosis of headache disorder other than chronic migraine (eg, cluster headache or medication overuse headache as per ICHD-IIIβ criteria24) or characterizes a pain disorder other than migraine as their primary presenting problem.
* Non-stable headache treatment regimen: Reports a change in physician prescribed preventive or acute headache pharmacotherapy within three weeks prior to enrollment or anticipates a change in preventive headache pharmacotherapy during the study period.
* Recent history of cardiovascular disease: Clinical history of cardiovascular disease (CVD) occurring within the past 6 months, including myocardial infarction, angina, coronary revascularization, stroke, TIA, carotid revascularization, peripheral arterial disease, and congestive heart failure. All persons with recent CVD should be participating in cardiac rehabilitation (with appropriate supervision as indicated) to reduce their risk of recurrence; hence, randomization might raise ethical concerns.
* Hypertension: Uncontrolled high blood pressure: BP > 160/100 mmHg. Potential participants can be re-screened after controlled.

Pregnancy, planning pregnancy and breast feeding (self-report) during screening: Pregnancy, breast feeding, or planning pregnancy within the next year.

* Physical preparedness for exercise: Those screening positive on the Physical Activity Readiness Questionnaire (PAR-Q)25 those must obtain physician clearance prior to participation, and will be excluded unless the clearance is obtained and documented.
* Other Medical and Psychiatric Conditions: Candidates will be screened for other co-morbid conditions that could make physical activity unsafe or limit participation. This includes other chronic disease likely to limit lifespan to less than 2-3 years (eg, any cancer requiring treatment in past 5 years except non-melanoma skin cancer), elevated depressive symptoms and/or suicidal ideation (Patient Health Questionnaire (PHQ-9)28,29), anxiety levels that could interfere with participation in this trial (PROMIS-29 Anxiety Subscale30-32, and evidence of opioid use disorder (Current Opioid Misuse Measure (COMM)33).
* Other: Conditions/criteria likely to interfere with participation and acceptance of randomized assignment, including the following: inability/unwillingness to give informed consent, another household member already randomized to HELP-VM, evidence of major psychiatric or cognitive problems (schizophrenia, dementia, self-reported active illegal substance or alcohol abuse), participation in another research study that would interfere with HELP-VM.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Acceptability- Number of participants recruited | 6 month
  To assess the acceptability of HELP-VM, the investigators will determine our ability to recruit Veterans to participate in the HELP-VM intervention as administered through the existing structure of the Salisbury VAMC's Whole Health Program
Percentage of adherence to HELP-VM | 6 month
  To evaluate the feasibility of implementing HELP-VM, the investigators will assess Veterans' adherence to HELP-VM
Number of participants that complete the intervention | 6 month
  To evaluate the feasibility of implementing HELP-VM, the investigators will assess our capacity to retain them in a clinical trial.
Mean of primary headache frequency | 6 month
  To evaluate the promise of HELP-VM, the investigators will obtain preliminary data to estimate variances (mean/SD) of primary headache frequency

CONTACTS AND LOCATIONS:
Overall Officials: Mara Vitolins, PhD, Principal Investigator — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: No